CLINICAL TRIAL: NCT06213415
Title: Role of Oral Steroid Alone Versus Oral Steroid Plus Intratympanic Steroid Injection in Bell's Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Alaa Abd-Alraheem, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Steroid injection bell's palsy
Record Dates: First submitted 2023-11-28; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Bell Palsy
MeSH Terms: conditions — Bell Palsy | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral steroids (Active Comparator): Oral steroids only
  Interventions: Drug: Corticosteroid
- Oral steroids plus intratympanic injections (Active Comparator): Oral steroids plus intratympanic injections
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Corticosteroid — Oral steroids plus intratympanic injection

SUMMARY:
intratympanic steroid injection bell's palsy

DETAILED DESCRIPTION:
Role of oral steroid alone versus oral steroid plus intratympanic steroid injection in Bell's palsy

ELIGIBILITY:
Inclusion Criteria:

* Mean Aged 18 years or more.

  * Acute unilateral facial palsy without skin lesions which developed within a 72-hour period and is present for 21 days or less.
  * Moderate to severe facial palsy [House-Brackmann grade IV or greater]

Exclusion Criteria:

* Another cause of facial nerve paralysis that is not idiopathic.

  * Otologic disease including otitis media, temporal bone fracture, a previous history of facial nerve palsy in either side, history of otologic surgery, and suspected Ramsay Hunt syndrome.
  * Systemic disease including history of tuberculosis, history of head and neck cancer, other neurological disorders, recent use of ototoxic medications, liver or renal dysfunction, and other illnesses that would contraindicate the use of high-dose steroid therapy.
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Success or failure of procedure to treat Bell's palsy | 6 months
  Degree of regaining function to facial nerve Unit of measurement : nerve conduction study
  Measurement tool :endoscopic injection by ear microscope

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ragab sayed, Study Director — Board membership

REFERENCES:
- [Background] Agostini F, Mangone M, Santilli V, Paoloni M, Bernetti A, Saggini R, Paolucci T. Idiopathic facial palsy: umbrella review of systematic reviews and meta-analyses. J Biol Regul Homeost Agents. 2020 Jul-Aug;34(4):1245-1255. doi: 10.23812/20-339-A. PMID 32935528
- [Background] Chang CWD, McCoul ED, Briggs SE, Guardiani EA, Durand ML, Hadlock TA, Hillel AT, Kattar N, Openshaw PJM, Osazuwa-Peters N, Poetker DM, Shin JJ, Chandrasekhar SS, Bradford CR, Brenner MJ. Corticosteroid Use in Otolaryngology: Current Considerations During the COVID-19 Era. Otolaryngol Head Neck Surg. 2022 Nov;167(5):803-820. doi: 10.1177/01945998211064275. Epub 2021 Dec 7. PMID 34874793
- [Background] Hernandez-Trejo AF, Cuellar-Calderon KP, Trevino-Gonzalez JL, Yamamoto-Ramos M, Campos-Coy MA, Quiroga-Garza A, Guzman-Avilan K, Elizondo-Riojas G, Elizondo-Omana RE, Guzman-Lopez S. Prevalence of facial canal dehiscence and other bone defects by computed tomography. Eur Arch Otorhinolaryngol. 2020 Oct;277(10):2681-2686. doi: 10.1007/s00405-020-06013-8. Epub 2020 May 7. PMID 32383094
- [Background] Inagaki A, Minakata T, Katsumi S, Murakami S. Concurrent Treatment With Intratympanic Dexamethasone for Moderate-Severe Through Severe Bell's Palsy. Otol Neurotol. 2019 Dec;40(10):e1018-e1023. doi: 10.1097/MAO.0000000000002377. PMID 31469789
- [Background] Volk GF, Schaede RA, Thielker J, Modersohn L, Mothes O, Nduka CC, Barth JM, Denzler J, Guntinas-Lichius O. Reliability of grading of facial palsy using a video tutorial with synchronous video recording. Laryngoscope. 2019 Oct;129(10):2274-2279. doi: 10.1002/lary.27739. Epub 2018 Dec 20. PMID 30570149
- [Background] Walker NR, Mistry RK, Mazzoni T. Facial Nerve Palsy. 2023 Jul 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK549815/ PMID 31747222